CLINICAL TRIAL: NCT01863498
Title: Prospective Randomized Trial: Pain Management After Pectus Excavatum Repair, Epidural Versus PCA
Brief Title: Prospective Trial: Pain Management After Pectus Excavatum Repair, Epidural Versus PCA
Acronym: PectusEpiPCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institution converted to an alternative strategy for pain control
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12120535
Record Dates: First submitted 2013-02-15; First posted 2013-05-29 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-08

CONDITIONS: Pectus Excavatum
Keywords: pectus excavatum; pain control
MeSH Terms: conditions — Funnel Chest; Agnosia | interventions — Injections, Epidural; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCA pain control (Active Comparator): Patients will have PCA for pain control
  Interventions: Other: PCA
- Epidural pain control (Active Comparator): Patients will have an epidural for pain control
  Interventions: Other: Epidural

INTERVENTIONS:
Other: Epidural — Patients will have an epidural for pain control
  Arms: Epidural pain control
Other: PCA — Patients will have PCA for pain control
  Arms: PCA pain control

SUMMARY:
Pectus excavatum, the most common chest wall deformity, occurs in roughly one in 1000 children. Operative repair of the anterior thoracic concavity has transitioned to the minimally invasive approach with substernal bar placement through small axillary incisions (Nuss procedure and multiple modifications). These procedures were quickly incorporated by high volume centers around the world including our own. The operation is certainly quicker and associated with less blood loss than the open operation, but as opposed to most minimally invasive versions of an operation, patients do not leave the hospital sooner after bar placement and experience more post-operative pain.

Pain during the post-operative hospital stay is the dominant management issue after bar placement. The sparse literature on the topic has suggested that a thoracic epidural is the most effective means for attenuating the pain during the first few post-operative days. Therefore, most centers approach all patients undergoing a pectus deformity repair with an attempt at epidural placement under the assumption that this provides the most effective strategy for pain control.

However, the investigators conducted a retrospective evaluation to examine the validity of this assumption and to investigate whether there is a role for a prospective study to determine the optimum post-operative pain management of these patients. The results demonstrate there was a decreased length of stay in the patients not treated with an epidural (PCA), despite no disadvantage in pain control. Further, 30% in whom an epidural was attempted, catheter placement failed.

This data certainly challenges the assumption that an epidural is the optimum management for these patients, and convincingly answers the question as to whether there is a role for a prospective randomized trial.

DETAILED DESCRIPTION:
Pectus excavatum, the most common chest wall deformity, occurs in roughly one in 1000 children.1 Operative repair of the anterior thoracic concavity has transitioned to the minimally invasive approach with substernal bar placement through small axillary incisions (Nuss procedure and multiple modifications). These procedures were quickly incorporated by high volume centers around the world including our own.2-7 The operation is certainly quicker and associated with less blood loss than the open operation, but as opposed to most minimally invasive versions of an operation, patients do not leave the hospital sooner after bar placement and experience more post-operative pain.6,7,8 Pain during the post-operative hospital stay is the dominant management issue after bar placement. The sparse literature on the topic has suggested that a thoracic epidural is the most effective means for attenuating the pain during the first few post-operative days.10-12 Therefore; most centers approach all patients undergoing a pectus deformity repair with an attempt at epidural placement under the assumption that this provides the most effective strategy for pain control.3-9, 13 However, the investigator conducted a retrospective evaluation to examine the validity of this assumption and to investigate whether there is a role for a prospective study to determine the optimum post-operative pain management of these patients.14 The investigator found length of stay was shorter with PCA and pain scores were similar. What the investigator found certainly challenges the assumption that an epidural is the optimum management for these patients, and convincingly answered the question as to whether there is a role for a prospective randomized trial.

The investigator conducted the prospective, randomized trial in 110 patients.15 The investigator found the pain scores were better with epidural for the first 2 days and better with PCA the last 2 days. There was no difference in length of stay although it trended to favor PCA. Epidural group incurred far greater operation times and charges. The pragmatic interpretation was that the investigator should just use PCA. The anesthesia interpretation is that the investigator need a better epidural. Therefore, the investigator have developed a better protocol for the transition to try to improve pain control the last 2 days. Further, the investigator recognize several flaws in the last study; the investigator included patients at extremes of age which don't represent a normal course. Second, the investigator kept patients in the hospital until they had a bowel movement which may have prolonged the care unnecessarily in the PCA group. The investigator will use the same sample size as last time since the difference in length of stay the investigator were designed to detect was more than a day which is clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a pectus excavatum repair with bar placement.
* Pectus patients between 12 and 17.9 years of age.

Exclusion Criteria:

* Open repair
* Re-Do operation
* Known allergy to a pain medication in the protocol
* Existing contraindications to epidural catheter placement
* Requirement for 2 bars to be placed (rare)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2013-05; Primary Completion 2018-01 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCA Pain Control | Epidural Pain Control
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCA Pain Control | Epidural Pain Control | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.3) | 15 (1.4) | 14.75 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 29 | 31 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: meters] | 1.8 (0.5) | 1.7 (0.1) | 1.75 (0.36)
Weight [Mean (Standard Deviation); unit: kg] | 53.9 (7.7) | 55.9 (10.4) | 54.88 (9.11)
Corrective Index [Mean (Standard Deviation); unit: index score] — Corrective Index scores of severity of pectus excavatum pre-surgery. Higher scores represent more severity. No minimum/maximum values. Scores on a scale.
  index score | 34.9 (9.6) | 28.6 (6.8) | 31.80 (8.86)

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization After Surgery
Description: The primary outcome variable is length of hospitalization after the intervention.
Time Frame: 3-8 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PCA Pain Control | Epidural Pain Control
Number analyzed (Participants) | 33 | 32
hours | 111.4 (51.4) | 111.3 (18.5)

2. Secondary Outcome: Operation Time
Description: Duration of operation in minutes
Time Frame: Duration of operation, an average of 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PCA Pain Control | Epidural Pain Control
Number analyzed (Participants) | 33 | 32
minutes | 58.9 (19.5) | 65.3 (22.9)

3. Secondary Outcome: Total Operating Room Time
Description: Total operating room time in minutes
Time Frame: Duration of time in operating room
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PCA Pain Control | Epidural Pain Control
Number analyzed (Participants) | 33 | 32
minutes | 102.8 (26.9) | 127.5 (28.4)

ADVERSE EVENTS:
Time Frame: From enrollment in trial until follow-up appointment, an average of 2 months
Arm/Group | PCA Pain Control | Epidural Pain Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT01863498/Prot_SAP_000.pdf